CLINICAL TRIAL: NCT04851041
Title: Long-term Effects of a Potato-based Food Pattern vs a Rice / Pasta-based Food Pattern on Fasting & Postprandial Cardiometabolic Health; The LoPoCardio - Trial
Brief Title: Effects of a Potato-based Food Pattern vs a Rice / Pasta-based Food Pattern on Cardiometabolic Health
Acronym: LoPoCardio
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: METC19-067
Record Dates: First submitted 2021-03-23; First posted 2021-04-20 (Actual); Last update posted 2021-04-20 (Actual); Status verified 2021-04

CONDITIONS: Glucose Metabolism; Lipid Metabolism
Keywords: Potato; pasta; rice; glucose metabolism; dietary patterns; Cardiometabolic health

STUDY DESIGN:
Intervention Model Description: Longer-term (12-weeks) well-controlled intervention trial with a parallel design including 56 overweight and obese (BMI25-35 kg/m2) men and women
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Potato group (Experimental): The participants in this group consume every day 150g of boiled potatoes for 12 weeks, preferably during dinner. The participants are allowed to eat this portion during lunch as well
  Interventions: Other: Potato
- Pasta/rice (Active Comparator): The participants in this group consume every day either rice or pasta for 12 weeks, preferably during dinner. The participants are allowed to eat this portion during lunch as well.
  The portion of rice and pasta must be as isocaloric as 150g of boiled potatoes.
  Interventions: Other: Pasta/rice

INTERVENTIONS:
Other: Potato — Controlled human intervention trial to evaluate the impact of boiled potato intake as part of a healthy dietary patterns on cardiometabolic health
  Arms: Potato group
Other: Pasta/rice — Since potatoes, white rice and white pasta are all products with a high glycemic index and concomitant relatively steep glucose excursions after intake, this intervention group helps to compare the effect of potato vs another high glucemic index food.
  Arms: Pasta/rice

SUMMARY:
The researchers investigate the effect of long-term (12-weeks) consumption of diets rich in boiled potatoes versus those rich in rice or pasta on established cardiovascular risk parameters. These carbohydrate sources will be part of a recommended healthy dietary pattern to mimic as closely as possible current dietary guidelines, facilitating the implementation of the outcomes.

DETAILED DESCRIPTION:
To breach the current controversies, there is an urgent need for well-designed controlled human intervention trials evaluating the true impact of boiled potato consumption as part of a healthy dietary pattern on cardiometabolic health. There are two important issues that need to be addressed when designing such an intervention study: First, the longer-term effects of boiled potato consumption on established fasting and postprandial cardiovascular risk markers should be addressed. Second, the effect of boiled potatoes should be studied using an iso-energetic exchange for other traditionally main carbohydrate sources. These carbohydrate-sources will be part of a recommended healthy dietary pattern to mimic as closely as possible current dietary guidelines, facilitating the implementation of the outcomes. Effects will be studied in both fasting and postprandial conditions. In fact, the evidence is accumulating that optimizing postprandial glucose and lipid responses are important targets for maintaining health. Since potatoes, white rice and white pasta are all products with a high glycemic index and concomitant relatively steep glucose excursions after intake, the question is how long-term intake of these products affects the metabolic capacity of our body to respond to postprandial challenges. Interestingly, potatoes are not only rich in complex carbohydrates but are also more nutrient-dense (a wide variety of minerals, vitamins, and micronutrients) as compared to white rice and white pasta. In addition, potatoes provide large amounts of fiber and are more satiating than other carbohydrate sources. This nutrient profile might beneficially impact the resilience of the metabolic machinery and as such improve postprandial cardiometabolic plasma profiles (glucose, insulin, and triacylglycerol). In other words, there might be a beneficial effect of longer-term potato consumption in comparison with longer-term white pasta and white rice consumption will not only be present in fasting conditions but particularly in the postprandial state when the cardiometabolic system is challenged.

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria are:
* Aged between 40-70 years
* Men and women
* 18-70 years
* BMI between 25-35 kg/m2 (overweight and obese)
* Serum total cholesterol < 8.0 mmol/L (further testing is recommended for excessive hyperlipidemia [serum total cholesterol ≥ 8.0 mmol/L] according to the Standard for cardiovascular risk management of the Dutch general practitioners community [NHG])
* Serum triacylglycerol < 4.5 mmol/L
* No current smoker
* No diabetic patients
* No familial hypercholesterolemia
* No abuse of drugs
* Not more than 4 alcoholic consumption per day with a maximum of 21 per week??
* Stable body weight (weight gain or loss < 3 kg in the past three months)
* No use of medication known to treat blood pressure, lipid or glucose metabolism
* No use of an investigational product within another biomedical intervention trial within the previous 1-month
* No severe medical conditions that might interfere with the study, such as epilepsy, asthma, kidney failure or renal insufficiency, chronic obstructive pulmonary disease, inflammatory bowel diseases, auto inflammatory diseases and rheumatoid arthritis
* No active cardiovascular disease like congestive heart failure or cardiovascular event, such as an acute myocardial infarction or cerebrovascular accident
* Willingness to give up being a blood donor from 8 weeks before the start of the study, during the study and for 4 weeks after completion of the study
* No difficult venipuncture as evidenced during the screening visit
* Willing to comply to study protocol during study
* Informed consent signed

Exclusion Criteria:

* The exclusion criteria are:
* Allergy or intolerance to potatoes, pasta or rice
* Serum total cholesterol ≥ 8.0 mmol/L
* Serum triacylglycerol ≥ 4.5 mmol/L
* Current smoker, or smoking cessation <12 months
* Diabetic patients
* Familial hypercholesterolemia
* Abuse of drugs
* More than 4 alcoholic consumptions per day or 21 per week
* Unstable body weight (weight gain or loss > 3 kg in the past three months)
* Use medication known to treat blood pressure, lipid or glucose metabolism
* Use of an investigational product within another biomedical intervention trial within the previous 1-month
* Severe medical conditions that might interfere with the study, such as epilepsy, asthma, kidney failure or renal insufficiency, chronic obstructive pulmonary disease, inflammatory bowel diseases, auto inflammatory diseases and rheumatoid arthritis
* Active cardiovascular disease like congestive heart failure or cardiovascular event, such as an acute myocardial infarction or cerebrovascular accident
* Not willing to give up being a blood donor from 8 weeks before the start of the study, during the study or for 4 weeks after completion of the study
* Not or difficult to venipuncture as evidenced during the screening visit
* Use of over-the-counter and prescribed medication or supplements, which may interfere with study measurements to be judged by the principal investigator;
* Use of oral antibiotics in 40 days or less prior to the start of the study;
* Blood donation in the past 3 months before the start of the study
* Not willing to comply to study protocol during study or sign informed consent

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2021-03-03 (Actual); Primary Completion 2024-05-01 (Estimated); Study Completion 2024-05-01 (Estimated)

PRIMARY OUTCOMES:
Chronic glucose metabolism | pre- intervention and post- intervention (12 weeks)
  Measured by change in average daily glucose concentrations over a 15 hours period between waking up and going to bed 7:00AM - 22:00PM for three days, which is calculated based on the total area under the curve (tAUC) using a continuos glucose monitor.

SECONDARY OUTCOMES:
Lipid metabolism | 12 weeks intervention: Pre-intervention (visit 1 and 2), during the intervention (visit 3, 4, 5) and post intervention (visit 6, and 7)
  Measured by fasting serum C-peptide, lipids and lipoproteins in all visits
Glucose metabolism | 12 weeks intervention: Pre-intervention (visit 1 and 2), during the intervention (visit 3, 4, 5) and post intervention (visit 6, and 7)
  Measured by fasting plasma glucose, insulin, and calculated HOMA- IR in all visits
Low grade inflammation | 12 weeks intervention: Pre-intervention (visit 1 and 2), during the intervention (visit 3, 4, 5) and post intervention (visit 6, and 7)
  Measured by inflammation plasma markers (hsCPR, IL6, IL8, TNFa)
Postprandial glucose metabolism | 12 weeks intervention: Pre-intervention (visit 2) and post intervention (visit 7)
  Following a high-fat, high-carb meal, measured by plasma glucose, insulin.
Postprandial TAG metabolism | 12 weeks intervention: Pre-intervention (visit 2) and post intervention (visit 7)
  Following a high-fat, high-carb meal, measured by plasma TAG.
24h urine samples micronutrient profiles | 12 weeks intervention: Pre-intervention (visit 2) and post intervention (visit 7)
  Measured by 24 urine collection.
Quality of life questionnaire | 12 weeks intervention: Pre-intervention (visit 2), during the intervention (visit 4) and post intervention (visit 7)
  Assessed with a 32-item questionnaire (including social, spiritual, emotional, cognitive, physical, activities of daily living, and integrated quality of life)
Mood, degree of pleasantness and arousal | 12 weeks intervention: Pre-intervention (visit 2), during the intervention (visit 4) and post intervention (visit 7)
  Assessed with the Affect grid
Fatigue | 12 weeks intervention: Pre-intervention (visit 2), during the intervention (visit 4) and post intervention (visit 7)
  Assessed using the FSS, a 9-item questionnaire that is used to determine the severity of fatigue a subject experienced in the past week during daily activities
Cognitive performance | 12 weeks intervention: Pre-intervention (visit 2), during the intervention (visit 4) and post intervention (visit 7)
  Assessed with a validated neuropsychological test battery (CANTAB)
Venular and arteriolar diameters | 12 weeks intervention: Pre-intervention (visit 2), during the intervention (visit 4) and post intervention (visit 7)
  Assessed via fundus photography
Office blood pressure | 12 weeks intervention: Pre-intervention (visit 1 and 2), during the intervention (visit 3, 4, 5) and post intervention (visit 6, and 7)
  Measured by office blood pressure monitor in all visits
36h blood pressure profiles | 12 weeks intervention: Pre- intervention (visit-1) and post- intervention (visit 6)
  Assessed via wearables blood pressure monitor

OTHER OUTCOMES:
Exploratory objective endothelial (dys)function markers | 12 weeks intervention: Pre-intervention (visit 1 and 2), during the intervention (visit 3, 4, 5) and post intervention (visit 6, and 7)
  Measured by sE-selectin, sICAM, sVCAM, and MCP-1 in al visits
  To investigate if potato consumption by overweight and obese (BMI25-35 kg/m2) men and women changes:
  * Endothelial (dys)function markers (sE-selectin, sICAM, sVCAM, and MCP-1) - Liver enzymes (e.g. ALAT, ASAT, gGT, bilirubin)
  * Calculated insulin secretory function (HOMA%B index)
  * Micro-albumineria and kidney function (estimated GFR)
  * Plasma incretins / satiety hormones (PYY, GLP, Ghrelin)
Exploratory objective liver enzymes | 12 weeks intervention: Pre-intervention (visit 1 and 2), during the intervention (visit 3, 4, 5) and post intervention (visit 6, and 7)
  Measured by liver enzymes (ALAT, ASAT, gGT, bilirubin)
Exploratory objective calculated insulin secretory function | 12 weeks intervention: Pre-intervention (visit 1 and 2), during the intervention (visit 3, 4, 5) and post intervention (visit 6, and 7)
  Measured by HOMA%B index
Exploratory objective micro-albumineria and kidney function | 12 weeks intervention: Pre-intervention (visit 1 and 2), during the intervention (visit 3, 4, 5) and post intervention (visit 6, and 7)
  Measured by estimated GFR
Exploratory objective plasma incretins / satiety hormones in fasting and postprandial conditions | 12 weeks intervention: Pre-intervention (visit 2) and post intervention (visit 7)
  Following a high-fat, high-carb meal, measured by PYY, GLP, ghrelin.

CONTACTS AND LOCATIONS:
Overall Officials: Jogchum J Plat, PhD, Principal Investigator — Chair of Nutrition and Movement Science Department; Ronald P. Mensisnk, PhD, Principal Investigator — Chair of Nutrition and Movement Science Department
Locations (1):
- Metabolic Research Unit Maastricht, Maastricht, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Seidelmann SB, Claggett B, Cheng S, Henglin M, Shah A, Steffen LM, Folsom AR, Rimm EB, Willett WC, Solomon SD. Dietary carbohydrate intake and mortality: a prospective cohort study and meta-analysis. Lancet Public Health. 2018 Sep;3(9):e419-e428. doi: 10.1016/S2468-2667(18)30135-X. Epub 2018 Aug 17. PMID 30122560
- [Background] Shan Z, Rehm CD, Rogers G, Ruan M, Wang DD, Hu FB, Mozaffarian D, Zhang FF, Bhupathiraju SN. Trends in Dietary Carbohydrate, Protein, and Fat Intake and Diet Quality Among US Adults, 1999-2016. JAMA. 2019 Sep 24;322(12):1178-1187. doi: 10.1001/jama.2019.13771. PMID 31550032
- [Background] Simpson SJ, Le Couteur DG, James DE, George J, Gunton JE, Solon-Biet SM, Raubenheimer D. The Geometric Framework for Nutrition as a tool in precision medicine. Nutr Healthy Aging. 2017 Dec 7;4(3):217-226. doi: 10.3233/NHA-170027. PMID 29276791
- [Background] Robertson TM, Alzaabi AZ, Robertson MD, Fielding BA. Starchy Carbohydrates in a Healthy Diet: The Role of the Humble Potato. Nutrients. 2018 Nov 14;10(11):1764. doi: 10.3390/nu10111764. PMID 30441846
- [Background] Jacome-Sosa M, Parks EJ, Bruno RS, Tasali E, Lewis GF, Schneeman BO, Rains TM. Postprandial Metabolism of Macronutrients and Cardiometabolic Risk: Recent Developments, Emerging Concepts, and Future Directions. Adv Nutr. 2016 Mar 15;7(2):364-74. doi: 10.3945/an.115.010397. Print 2016 Mar. PMID 26980820
- [Background] King JC, Slavin JL. White potatoes, human health, and dietary guidance. Adv Nutr. 2013 May 1;4(3):393S-401S. doi: 10.3945/an.112.003525. PMID 23674809
- [Background] Camire ME, Kubow S, Donnelly DJ. Potatoes and human health. Crit Rev Food Sci Nutr. 2009 Nov;49(10):823-40. doi: 10.1080/10408390903041996. PMID 19960391